CLINICAL TRIAL: NCT04770064
Title: Targeting Senescence to Reduce Osteoarthritis Pain and cartilagE Breakdown (ROPE)
Acronym: ROPE
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Funding was not awarded
Sponsor: Austin V Stone (Other)
Collaborators: Brigham and Women's Hospital (Other)
Responsible Party: Sponsor-Investigator, Austin V Stone, Assistant Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 65448
Record Dates: First submitted 2021-02-16; First posted 2021-02-25 (Actual); Last update posted 2022-07-29 (Actual); Status verified 2022-07

CONDITIONS: Osteoarthritis, Knee
Keywords: Knee; Osteoarthritis; Pain; Inflammation
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis; Pain; Inflammation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- High-dose/short-duration Fisetin (FIS-hi) (Experimental)
  Interventions: Drug: High-dose/short-duration Fisetin
- Low-dose/sustained duration Fisetin (FIS-lo) (Experimental)
  Interventions: Drug: Low-dose/sustained-duration Fisetin
- Placebo (Placebo Comparator)
  Interventions: Other: Oral placebo capsule

INTERVENTIONS:
Drug: High-dose/short-duration Fisetin — Fisetin is a plant flavanol senolytic found in strawberries, persimmons, and cucumbers. It has senolytic properties that may provide therapeutic benefit for those with knee osteoarthritis. Participants will be asked to take approximately 20 mg/kg of body mass for 2 consecutive days, followed by a 28-day washout period, and then another 2-day administration.
  Arms: High-dose/short-duration Fisetin (FIS-hi)
Drug: Low-dose/sustained-duration Fisetin — Fisetin is a plant flavanol senolytic found in strawberries, persimmons, and cucumbers. It has senolytic properties that may provide therapeutic benefit for those with knee osteoarthritis. Participants will be asked to take one, 100 mg capsule of fisetin daily for 90 days.
  Arms: Low-dose/sustained duration Fisetin (FIS-lo)
Other: Oral placebo capsule — Participants will be asked to take one, 100 mg oral placebo capsule (corn starch) daily for 90 days.
  Arms: Placebo

SUMMARY:
Symptomatic knee osteoarthritis (OA) is the most common joint disorder in the U.S. and a leading cause of disability. Increasing age, obesity, and previous injury increase the lifetime risk of knee OA, but these factors are also independently associated with increased cellular senescence. Senescent cells accumulate in many tissues and contribute to chronic pathologies, linked to the secretion of pro-inflammatory factors collectively known as the senescence-associated secretory phenotype. In OA, senescent cells promote production of cytokines, chemokines, and matrix-degrading enzymes involved in progressive cartilage breakdown. The senolytic supplement fisetin alters the inflammatory and catabolic cartilage responses, which may clinically lessen OA pain while also slowing progressive cartilage breakdown. The purpose of this double-blind, randomized clinical trial is to compare 2 fisetin dosing regimens versus placebo. Sixty patients with mild to moderate knee OA will be assessed at baseline and 3 months in an effort to: determine if 2 different fisetin dosing regimens lessen pain and functional impairment compared to placebo, compare progressive changes in senescent cell activity and biomarkers of cartilage degradation between different fisetin dosing regimens and placebo, and assess acceptability and feasibility of 2 fisetin dosing regimens.

ELIGIBILITY:
Inclusion Criteria:

* Are male or female, ages 35-80;
* Are willing to comply with all study related procedures and assessments;
* Are ambulatory as defined by ability to complete functional performance testing;
* Radiographic evidence of Kellgren-Lawrence grade II-IV osteoarthritis in one or both knees;
* Scores between 40 and 80 mm on the pain VAS;
* Stable dose of screening/baseline medications for at least 2 months prior to the anticipated date of study drug dosing.

Exclusion Criteria:

* Females who are nursing, pregnant or planning to become pregnant during the duration of study drug dosing;
* Males who do not wish to abstain from sex or use contraceptive protection during study drug dosing and for 2 weeks after the last dose;
* Subjects who do not have the capacity to consent themselves;
* Subjects who are unable to tolerate oral medication;
* Subjects having previously undergone any of the following treatments in the stated time window.
* Surgery on the Study Knee in the past 6 months;
* Partial or complete joint replacement in the study knee. Partial or complete joint replacement in the contralateral knee is acceptable as long as the surgery was performed at least 6 months prior to enrollment and the operative knee is asymptomatic;
* Patients who have undergone arthroscopic surgery (including microfracture and meniscectomy) on the Study Knee in the last 2 years prior to the Screening visit or are anticipated to have arthroscopic surgery on either knee at any time during the study period;
* Patients that have had a recent intraarticular OA treatment:
* Glucocorticoid injection, within the last 2 months;
* Extended-release corticosteroid, hyaluronic acid, or biologic injection (platelet-rich plasma, bone marrow, adipose tissue/cells) into the Study Knee in the past 6 months;
* Subjects with any of the following drug/medication statuses:
* Currently taking Losartan;
* Currently taking Warfarin or related anticoagulants;
* Opioid analgesics taken in the past 8 weeks;
* Senolytic agents taken within the past 6 months and are not willing to discontinue these medications through the duration of the study, including: Fisetin, Quercetin, Luteolin, Dasatinib, Piperlongumine, or Navitoclax;
* Drugs that induce significant cellular stress and are not willing to discontinue these medications through the duration of the study, including alkylating agents, anthracyclines, platins, other chemotherapy drugs;
* Subjects taking the following other drugs if they cannot be held (per the Principal Investigator) for at least 2 days before and during administration of Fisetin: cyclosporine, tacrolimus, repaglinide, and bosentan.
* Subjects with any of the following disease statuses:
* Significant liver disease (i.e. greater than or equal to 2x the upper limit of normal bilirubin levels) or as in the opinion of the Principal Investigator;
* Significant renal disease (eGFR of <60 ml/min/1.73m2) or as in the opinion of the Principal Investigator;
* History of other formally diagnosed joint diseases including osteonecrosis, acromegaly, Paget's disease, Ehlers-Danlos Syndrome, Gaucher's disease, Cushing's syndrome, Stickler's syndrome, joint infection, hemophilia, hemochromatosis, or neuropathic arthropathy of any cause;
* Any active systemic autoimmune disease with musculoskeletal involvement or any history of system inflammatory arthritis;
* Patients with type 1 or 2 diabetes (HbA1c>6.5%) and/or taking medications that affect insulin levels, including: Metformin (within the last week), Glucocorticoids (within the last month), Acarbose (within the last week);
* Subjects with moderate to severe depression (PHQ-9 score > 10) will also be excluded since knee OA patients with depression have previously demonstrated worse pain trajectories;
* Subjects that have any medical condition, including laboratory findings and findings in the medical history or in the pre-study assessments, that in the opinion of the Investigator constitutes a risk or contraindication for participation in the study or that could interfere with the study objectives, conduct or evaluation or prevent the patient from fully participating in all aspects of the study.

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-06 (Estimated); Primary Completion 2024-05-31 (Estimated); Study Completion 2024-05-31 (Estimated)

PRIMARY OUTCOMES:
Change in markers of liver toxicity | Change between baseline and 3-month follow-up
  The change in 2 markers of liver toxicity between baseline and 3-month follow-up will be assessed. Alanine amino transferase (ALT) and aspartate amino transferase (AST) are enzymes found mostly in the cells of the liver and kidney, and heart and liver, respectively. Both are useful tests for detecting liver damage.
Change in markers of kidney toxicity | Change between baseline and 3-month follow-up
  The change in 2 markers of kidney toxicity between baseline and 3-month follow-up will be assessed. Blood urea nitrogen (BUN) is a waste product filtered out of the blood by the kidneys. As kidney function decreases, the BUN level rises. Creatine kinase (CK) is also an enzyme that is used to assess kidney function. Higher CK values are associated with greater burden on the kidneys.
Change in markers of tumor lysis syndrome | Change between baseline and 3-month follow-up
  Tumor lysis syndrome is characterized by high blood potassium, low blood calcium, and high blood uric acid. The change in potassium, calcium and uric acid between baseline and 3-month follow-up will be assessed.

SECONDARY OUTCOMES:
Pain Visual Analogue Scale (VAS) | Change between baseline and 3-month follow-up
  The Pain VAS is a 100 mm scale where participants will be asked to report their level of pain over the past 24 hours, with 0 being associated with no pain and 100 mm being associated with the worst pain imaginable.
Western Ontario and MacMaster Universities Osteoarthritis Index (WOMAC) | Change between baseline and 3-month follow-up
  The WOMAC is a 24-item instrument that has been found to be valid and responsive when quantifying changes in pain and function in individuals with knee osteoarthritis. Scores range from 0 to 96 with higher WOMAC scores being associated with worse pain, stiffness, and functional limitations.
Five times sit-to-stand test | Change between baseline and 3-month follow-up
  The five-repetition sit-to-stand is commonly used to measure mobility and function in older adults. Participants are positioned in a standard 16" office chair with their arms at their sides and back located against the back of the chair. Participants are instructed to "Please stand up straight as quickly as you can 5 times, without stopping in between. Keep your arms folded across your chest. I'll be timing you with a stopwatch. Ready, begin." The test is timed using a stopwatch and the timer is stopped when the individual achieves a standing position on the 5th trial. Faster times are associated with less functional impairment.
Biomarker of cellular senescence (MMP-3) | Change between baseline and 3-month follow-up
  Matrix metalloproteinase-3 (MMP-3) is commonly associated with senescence-associated secretory phenotype, and have been previously used to assess the mechanism of action of fisetin in human clinical trials. Greater serum concentrations of MMP-3 are associated with increased senescent cell activity.
Biomarker of cartilage breakdown (CTXII) | Change between baseline and 3-month follow-up
  C-terminal crosslinked telopeptide type II collagen (CTXII) has been identified as a biomarker for the diagnosis, staging, and evaluating the prognosis of hip and knee osteoarthritis, and has also been demonstrated to be responsive over short testing periods (3 months). Greater concentrations are associated with increased cartilage breakdown. CTXII will be measured in the urine and will be normalized to creatinine levels.

OTHER OUTCOMES:
Need for rescue treatment | 3-month follow-up
  We will record the prevalence and time to rescue intra-articular injections such as a corticosteroid injection.
Treatment Adherence | 3-month follow-up
  Participants will be asked to complete an adherence questionnaire weekly throughout the study period. Participants will be contacted via their preferred method (phone, email, SMS text message). Previous literature has defined good medication compliance as taking at least 80% of the prescribed medication. We will calculate the proportion of patients who meet this criterion in the treatment group as well as the 95% confidence interval (CI) around this compliance rate. The treatments will be considered feasible and acceptable if over 70% of participants reach this threshold.

CONTACTS AND LOCATIONS:
Overall Officials: Austin Stone, MD, PhD, Principal Investigator — University of Kentucky
Locations (2):
- United States (2):
  - UK Healthcare at Turfland, Lexington, Kentucky
  - UK HealthCare Joint Reconstruction and Replacement, Lexington, Kentucky

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IDP) will not be made available to other researchers.